CLINICAL TRIAL: NCT04627493
Title: Improving Physical Activity and Mobility, During a Pandemic, Via Live Online Exercise Sessions for Older Persons: a Pilot RCT
Brief Title: Improving Physical Activity and Mobility Via Live Online Exercise Sessions for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11429
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Aging
Keywords: Exercise; Online
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will be a randomized parallel-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist (Control) (No Intervention): Usual care
- Exercise (Experimental): Online exercise program
  Interventions: Behavioral: Online exercise

INTERVENTIONS:
Behavioral: Online exercise — Participants will participate in an online exercise program on Zoom delivered by Registered Kinesiologists and Physiotherapists three times a week.
  Arms: Exercise

SUMMARY:
The COVID-19 pandemic has undoubtedly resulted in an increased level of personal anxiety, reduced access to support services, and as a secondary complication, increased physical inactivity. Older people appear to be at higher risk of several secondary complications and long-term negative health outcomes. These complications include declines in physical health and mobility, social isolation, and worsening mental health. There is strong evidence in older persons that supports the role of exercise and physical activity in: the alleviation of strength and mobility declines, reducing anxiety and depression, and alleviating cognitive declines. Exercise-based intervention trials have also been shown to reduce social isolation and loneliness. This study will compare an online exercise program delivered via Zoom and a waitlist control group in healthy older persons.

DETAILED DESCRIPTION:
This study will examine the impacts of an online exercise program in healthy older persons compared to a waitlist control group. Briefly, participants (healthy persons, age 65-80 years old) will participate in an online group exercise program (designed to meet Canada's Physical Activity Guidelines) via Zoom delivered by Registered Kinesiologists and Physiotherapists for a total of 8 weeks. Participants will be randomly assigned to the exercise group or the waitlist control group. Participants' will undergo assessments of physical activity, life-space mobility, nutrition, loneliness, depression, and anxiety at baseline, end of study, and 8-weeks following the end of the intervention.

ELIGIBILITY:
Exclusion Criteria:

1. Experience any physical conditions which may prevent them from engaging in moderate-intensity physical activity including using assistive walking devices (e.g. cane or walker), or injuries;
2. Have a history of neuromuscular conditions or muscle wasting diseases;
3. Are currently participating in physical activity, ≥150 minutes of moderate-to-vigorous physical activity per week;
4. Are not eligible to participate in regular physical activity according to the Canadian Society Exercise Physiology Get Active Questionnaire;
5. Do not have access to the internet at home via a personal smartphone, tablet (e.g., iPad), or computer.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Changes in physical activity | Baseline, post intervention, 8-week follow-up
  7 day steps and activity-related energy expenditure

SECONDARY OUTCOMES:
Change in life-space mobility score | Baseline, post intervention, 8-week follow-up
  The University of Alabama Life Space Assessment, UA-LSA, will be used to assess participants life-space mobility score. It is a global marker of older adults' physical and community mobility and it has been shown to relate to objectively-measured step counts.
Change in nutrition | Baseline, post intervention, 8-week follow-up
  The Screen II (Seniors in the Community Risk Evaluation for Eating and Nutrition) will be used to determine whether individuals have a potential nutritional problem or are at risk of developing one and identifies those who need further nutrition assessment and treatment.
Change in feelings of loneliness | Baseline, post intervention, 8-week follow-up
  The 11-item Revised University of California Los Angeles loneliness scale (R-UCLA) will be used to assess participants' feelings of loneliness.
Change in the Geriatric Depression Scale score | Baseline, post intervention, 8-week follow-up
  The Geriatric Depression Scale (GDS-15) contains 15 items that measure the intensity of depressive symptoms on a dichotomous scale (yes or no). The total score ranges from 0 to 15. Higher scores indicate higher levels of depressive symptoms.
Change in the Geriatric Anxiety Inventory score | Baseline, post intervention, 8-week follow-up
  The Geriatric Anxiety Inventory (GAI) contains 20 items that measure the intensity of anxious symptoms on a dichotomous scale (agree or disagree). The total score ranges from 0 to 20. A score of 10 or over is associated with the presence of a generalized anxiety disorder (GAD).
Program Feasibility | Throughout the participant's intervention period (0-8 weeks)
  Program feasibility will be evaluated by: 1) program adherence/attendance in the online exercise program for participants in the intervention group; and 2) program satisfaction/acceptability questionnaire at the end of each online exercise class for all participants in the intervention group.
Participants experiences and perceptions | 1-60 days post intervention
  Participants' experiences and perceptions of exercise and our online exercise program. This will be collected through qualitative data: semi-structured one-on-one interviews conducted with each participant who completes the online exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University
Locations (1):
- Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coletta G, Noguchi KS, Beaudoin KD, McQuarrie A, Tang A, Griffin M, Ganann R, Phillips SM. A live online exercise program for older adults improves depression and life-space mobility: A mixed-methods pilot randomized controlled trial. PLoS One. 2024 Nov 11;19(11):e0312992. doi: 10.1371/journal.pone.0312992. eCollection 2024. PMID 39527532